CLINICAL TRIAL: NCT01548105
Title: Systemic Markers of Collagen Metabolism and Vitamin C in Smokers and Non-Smokers With Pelvic Organ Prolapse
Status: Completed | Type: Observational
Sponsor: TriHealth Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: Smoking and prolapse
Record Dates: First submitted 2012-03-04; First posted 2012-03-08 (Estimated); Last update posted 2014-10-17 (Estimated); Status verified 2014-02

CONDITIONS: Pelvic Organ Prolapse
Keywords: Pelvic organ prolapse; smoking and collagen metabolism
MeSH Terms: conditions — Pelvic Organ Prolapse; Smoking | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Prolapse and Smoker: Patients in this arm have been determined to have more than stage 2 pelvic organ prolapse and have been smoking more than one pack per day Blood draw for the study participants will be done. These will include: Procollagen 1-N propeptide levels (PINP), Matrix metalloproteinase (MMP9) and Plasma Vitamin C levels
  Interventions: Other: Blood draw for the study participants
- Prolapse and non smoker: Patients in this arm have been determined to have more than stage 2 pelvic organ prolapse and non smoker for more than 7 years Blood draw for the study participants will be done. These will include: Procollagen 1-N propeptide levels (PINP), Matrix metalloproteinase (MMP9) and Plasma Vitamin C levels
  Interventions: Other: Blood draw for the study participants
- No prolapse and smoker: Patients in this arm, have been determined not to have prolapse and smokes more than 1 pack per day Blood draw for the study participants will be done. These will include: Procollagen 1-N propeptide levels (PINP), Matrix metalloproteinase (MMP9) and Plasma Vitamin C levels
  Interventions: Other: Blood draw for the study participants
- No prolapse and non smoker: Patients in this arm have been determined not to have prolapse and non smoker for more than 7 years Blood draw for the study participants will be done. These will include: Procollagen 1-N propeptide levels (PINP), Matrix metalloproteinase (MMP9) and Plasma Vitamin C levels
  Interventions: Other: Blood draw for the study participants

INTERVENTIONS:
Other: Blood draw for the study participants — These will include:
  * Procollagen 1-N propeptide levels (PINP)
  * Matrix metalloproteinase (MMP9)
  * Plasma Vitamin C levels

SUMMARY:
Data on smoking and POP are conflicting. In a study done by Alnaif et al, smoking was found to be associated with severe POP. The authors' proposed explanation was that smoking impairs tissue and wound healing. Our primary objective is to document whether smokers with pelvic organ prolapse (POP) are different from non-smokers with POP with respect to collagen biosynthesis and breakdown using systemic markers of collagen metabolism and Vitamin C.

DETAILED DESCRIPTION:
Tissue destructive disorders are more common in smokers than in non-smokers. Alterations in wound healing and connective tissue turnover are suggested mechanisms, but exact details remain to be discovered. The synthesis of subcutaneous collagen in smokers is specifically impeded, and that smokers have less collagen compared to non-smokers. Jorgensen et al study showed that smokers tend to have less procollagen I N-propeptide (PINP) levels in the blood, less vitamin C and higher levels of matrix metalloproteinase (MMP-9), these findings reversed after smoking cessation.

Since smoking is one of the promoting and modifiable factors in the development of prolapse, understanding its effects on the support of pelvic organs may help modify the course of the POP condition in the future. Understanding the connective tissue effects of smoking using systemic markers of collagen metabolism in female smokers with prolapse may help future management and counseling of these patients. In addition, description of the markers of collagen metabolism in POP has not previously been documented.

ELIGIBILITY:
Inclusion Criteria: PROLAPSE group

* More than 18 years old
* Symptomatic POP at or beyond the hymen as determined by physical examination and a positive answer to the screening questions
* For smoker group- smoke more than one pack per day
* For non smoker group- non smoker for more than 7 years

No Prolapse group:

* Absence of prolapse and negative answer to the screening questions

Exclusion Criteria:

* Using Hormone Replacement Therapy (systemic estrogen, progesterone or testosterone)
* Using vaginal estrogen (cream, ring, tablet)
* Chronic steroid use
* Past medical history of connective tissue disease
* Scurvy, malabsorption, alcoholism, pregnancy, hyperthyroidism, liver disease and renal failure

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with pelvic organ prolapse and without prolapse will be identified based on a manual review of patients in a tertiary care referral-based Urogynecology practice
Sampling Method: Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2012-03; Primary Completion 2013-01 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Our primary objective is to document whether smokers with pelvic organ prolapse (POP) are different from non-smokers with POP with respect to collagen biosynthesis and breakdown using systemic markers of collagen metabolism. | One day- day of blood draw
  These will include blood levels of the following:
  * Procollagen 1-N propeptide levels (PINP)
  * Matrix metalloproteinase (MMP9)
  * Plasma Vitamin C levels

SECONDARY OUTCOMES:
• A secondary objective will be to determine whether women with pelvic organ prolapse are different than healthy controls with respect to the same systemic markers | One day- day of blood draw

CONTACTS AND LOCATIONS:
Overall Officials: Maria Victoria C Estanol, MD, Principal Investigator — Good Samaritan Hospital
Locations (1):
- Good Samaritan Hospital, Cincinnati, Ohio, United States